CLINICAL TRIAL: NCT01612026
Title: Ultrasound Versus Fluoroscopically-guided Arterial Access in Non-cardiac Vascular Patients
Status: Completed | Type: Observational
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Patrick Stone, MD, Study Principal Investigator, CAMC Health System
Other Study IDs: 1997155
Record Dates: First submitted 2012-05-23; First posted 2012-06-05 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2019-05

CONDITIONS: Arterial Cannulation During Vascular Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ultrasound
  Interventions: Procedure: arterial cannulation by angiographic imaging
- Fluoroscopy
  Interventions: Procedure: arterial cannulation by angiographic imaging

INTERVENTIONS:
Procedure: arterial cannulation by angiographic imaging — comparing successful arterial cannulation in case of non-cardiac vascular patient population.

SUMMARY:
In the investigators vascular practice, either fluoroscopic- or ultrasound-guided technique is routinely used to obtain femoral arterial access. Ultrasound-guidance is frequently used in patients with weak or absent pulses, known abnormal vascular anatomy, need for bypass graft puncture, and to ensure accurate arterial puncture in patients expected to receive large doses of blood-thinning medications during or after the procedure. For those practitioners experienced with ultrasound-guided access techniques, it is considered highly accurate and easy to use; thus, some physicians routinely use this tool. A well-designed study is needed to truly assess the accuracy of the ultrasound technique and to determine whether it may reduce complications of arterial access in vascular patients.

By demonstrating the safest, most accurate and efficient technique for obtaining arterial access during catheter-based procedures, the investigators could significantly reduce morbidity and mortality associated with complications of arterial puncture. Length of hospital stay, management costs and patient discomfort could be reduced by minimizing complication rates.

DETAILED DESCRIPTION:
Arterial access accounts for the highest frequency of complications in catheter-based procedures in the U.S. In our vascular practice, ultrasound-guidance is frequently used in patients with weak or absent pulses, known aberrant vascular anatomy, need for graft puncture, and to ensure accurate arterial puncture in patients expected to receive large doses of anti-thrombotic medications. Some practitioners routinely use this modality. The purpose of this study is to determine whether real-time ultrasound guidance is superior to fluoroscopic guidance in obtaining successful arterial cannulation during diagnostic and interventional catheter-based procedures in a primarily non-cardiac vascular patient population. Patients will be randomized to receive either real-time ultrasound-guided arterial access or fluoroscopic-guided access. Baseline patient demographics, co-morbidities, medications, pertinent laboratory data, and indications for procedure will be recorded. Procedural data recorded will include procedure type, type of access, operator, pulse quality, sheath size, closure device, angiographic data for access artery, antithrombotic medications used, and intra-procedural activated clotting times. Primary endpoint will be successful arterial cannulation by angiographic imaging. Secondary end points will be time to access, number of attempts, accidental venipunctures, first pass success, complication rates and hospital length of stay. Data regarding complications (patient history, examination, laboratory or imaging studies) will be included for a period of 90 days after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years of age undergoing a non-cardiac catheter-based diagnostic or interventional procedure requiring femoral artery cannulation. This will include patients with co-morbid conditions of coronary artery disease and other cardiac health problems.

Exclusion Criteria:

1. Patients less than 18 years of age.
2. Patients enrolled in another IRB approved biomedical study.
3. Pregnant females.
4. Prisoners.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects referred to the West Virginia University Department of Surgery: Division of Vascular and Endovascular Surgery with accepted indications to undergo a catheter-based diagnostic or interventional procedure requiring arterial cannulation.Procedures include peripheral, renal, mesenteric and carotid.
Sampling Method: Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of successful arterial cannulation by ultrasound and by fluoroscopy i.e. between two groups. | within 30 days

SECONDARY OUTCOMES:
Number of attempts, accidental venipunctures, first pass success, complications for arterial cannulation by ultrasound and by fluoroscopy i.e. between two groups. | within 30 to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stone, M.D., Principal Investigator — CAMC Medical Staff-with admitting privileges
Locations (1):
- Vascular Center of Excellence, Charleston, West Virginia, United States

REFERENCES:
- [Result] Stone P, Campbell J, Thompson S, Walker J. A prospective, randomized study comparing ultrasound versus fluoroscopic guided femoral arterial access in noncardiac vascular patients. J Vasc Surg. 2020 Jul;72(1):259-267. doi: 10.1016/j.jvs.2019.09.051. Epub 2020 Jan 21. PMID 31980242